CLINICAL TRIAL: NCT03451032
Title: Regional Multicenter Study to Evaluate Tolerability and Efficacy of TAF/FTC/RPV Combination (ODEFSEY ®) in Prevention of Sexual or Blood Exposure to HIV
Acronym: AES ODEFSEY
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0485
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hiv
Keywords: HIV exposition treatment; sexual risk; blood risk
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non Interventional Study — Non Interventional Study

SUMMARY:
Prospective, multicenter study to evaluate tolerability, adherence and efficacy of a 28-day course of TAF/FTC/RPV, an HIV post-exposure prophylaxis after a potential sexual or blood exposure to HIV.

At baseline, participants are prescribed TAF/FTC/RPV and a blood test. At W6, all participants are contacted by phone to evaluate completeness and tolerability of the TAF/FTC/RPV regimen.

DETAILED DESCRIPTION:
At baseline, participants seek care in one of the centers of " Pays de la Loire " area after a potential HIV exposure. They receive TAF/FTC/RPV, one pill taken with food once daily for 28 days according to national guidelines. They have to start this post-exposure prophylaxis within 48 hours after the HIV exposure.

At inclusion, participants give their written consent to have their data recorded in an electronic medical record Nadis® and their oral consent after reading the study information letter. A blood test is prescribed to examine biological variables (HIV, HBV, HCV serologies, TPHA VDRL, ALT/AST, hemogram and serum creatinine). Characteristics of participants and context of the risk are collected in the electronic medical record Nadis®. A blood test is prescribed at W2, W6 and W12 to evaluate tolerability and efficacy of the treatment.

At W6, all participants are contacted by phone call to evaluate completeness and tolerability of the TAF/FTC/RPV regimen. They are reminded to have a blood test done at W6 and W12.

ELIGIBILITY:
Inclusion Criteria:

* Subject seeking care in one of the French CEGIDD or in one of the French centers of " Pays de la Loire " area (CHU Nantes, CHU Angers, CHD La Roche sur Yon, CH Le Mans, CH Saint Nazaire, CH Laval) after a potential sexual or non-sexual HIV exposure
* Adult ≥18 years old
* Oral informed consent
* Written informed consent to have their data recorded in an electronic medical record ("Nadis" software).
* Indication of HIV post-exposure prophylaxis according to the French guidelines

Exclusion Criteria:

* Subject not willing or refusing to participate
* Subject on legal protection
* HIV positive status
* Pregnancy or breastfeeding
* Already treated by pre exposure prophylaxis
* Already included in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons included in the study are adults who seek care in one of the French CEGIDD or in one of the French centers of " Pays de la Loire " area after a potential sexual or blood HIV exposure with an indication of HIV post-exposure prophylaxis according to the French guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who stopped the 28-day course of TAF/FTC/RPV | At 6 weeks
  : Phone call to all participants to check on their adherence and to collect information about possible side effects

SECONDARY OUTCOMES:
Proportion of participants who had side effects of the post-exposure prophylaxis with TAF/FTC/RPV | At 6 weeks
  Phone call to all participants to collect information about possible side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte BONNET, Dr, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Laval Hospital, Laval
  - Le Mans Hospital, Le Mans
  - Nantes University Hospital, Nantes
  - Saint-Nazaire Hospital, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No